CLINICAL TRIAL: NCT03889028
Title: Pre-engraftment Cytomegalovirus DNAemia in Allogeneic Hematopoietic Stem Cell Transplant Recipients: Incidence, Risk Factors and Clinical Outcomes
Brief Title: Pre-engraftment Cytomegalovirus DNAemia
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, David Navarro, David Navarro, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: NAV-CMV-2019
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: CMV DNAemia Pre-engraftment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cytomegalovirus (CMV) DNAemia occurs frequently in allogeneic hematopoietic stem cell transplant (allo-HSCT) recipients.Both high-level and persistent virus DNAemia are known risk factors for CMV end-organ disease and perhaps non-relapse mortality. CMV DNAemia is usually documented after engraftment, but it may occur before. The virological features and clinical consequences of these latter early-onset episodes remain largely unexplored. The U.S. Food and Drug Administration (FDA) has recently approved letermovir for prophylaxis of CMV infection and disease in adult CMV-seropositive allo-HSCT recipients (PREVYMIS™, Merck & Co., New Jersey, USA). In accordance with the design of the phase III, double-blind trial the drug may be administered as early as the day of transplant and no later than 28 days post-transplant. Nevertheless, the timing of drug inception should be contingent on the clinical impact of very early episodes of CMV DNAemia. In a recent work from our group (single-center study) we found that a total 38 out of the 197 patients in our series developed CMV DNAemia before engraftment (cumulative incidence (CI), 19%; 95% CI, 10-30.3%). Nine episodes of CMV DNAemia were detected prior to the time of donor progenitor cell infusion. A greater number of post-engraftment episodes required preemptive antiviral therapy compared with pre-engraftment episodes (62.5% vs 44.7%; P=0.05). The cellular content of the donor progenitor cell infusion and transplant characteristics of patients did not differ between patients with pre- or post-engraftment CMV DNAemia. The cumulative incidence of overall mortality by days 100 and 365, aGvHD by day 100 and relapse by day 365 were not significantly different between patients with pre-engraftment or post-engraftment CMV DNAemia. Our study was limited by the retrospective and single-center design and the scarce number of pre-engraftment CMV DNAemia episodes included; therefore, the results may not be extrapolated to other transplantation centers or patient cohorts. Further retrospective and prospective studies are thus required to validate the data presented herein.

DETAILED DESCRIPTION:
Episodes of CMV DNAemia developing prior to engraftment (pre-CMV DNAemia), which usually occur between the third and fourth week after allo-HSCT, may conceivably have a different course from episodes emerging after engraftment once patients have begun to expand donor-derived T cells (post-CMV DNAemia). Thus, whether the precise timing of Letermovir treatment initiation should matter will ultimately depend on the impact of CMV DNAemia episodes developing prior to engraftment on clinical outcomes. There is limited information available on this topic. Here, we conducted a retrospective multicenter, non-interventional study to further address this issue.

ELIGIBILITY:
Inclusion Criteria:

* Recipients >18 years old
* CMV seropositive recipients and/or donors
* First allo-HSCT (T cell replete)
* CMV DNA load monitoring by real-time PCR

Exclusion Criteria:

* Recipients < 18 years
* CMV seronegative donors and recipients.
* No CMV DNA load monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive allo-HSCT recipients at risk of CMV infection allografted from 1st January 2010 until 31th December 2017 in Spanish transplant centers
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical University Hospital of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients undergoing T-cell replete allo-HSCT at 20 different centers in Spain from September 2014 to December 2015 (Registry of the Working group on Infectious and Non-Infectious Complications of the GETH-Spanish Hematopoietic Transplantation and Cell Therapy Group-). A total of 218 adult patients who received an unmanipulated allo-HSCT at the Clinical University Hospital of Valencia from March 2010 to May 2019 (excluding patients recruited in the GETH registry) were also included
Units Other Than Participants: Patients with or without CMV DNAemia
Groups:
- Pre-CMV DNAemia: Patients who developed CMV DNAemia prior to engraftment
- Post-CMV DNAemia: Patients with CMV DNAemia detected after neutrophil's engraftment
- No CMV DNAemia: Patients without CMV DNAemia throughout the study period
Period: Overall Study
Arm/Group | Pre-CMV DNAemia | Post-CMV DNAemia | No CMV DNAemia
Started | 144; 144 Patients with or without CMV DNAemia | 422; 422 Patients with or without CMV DNAemia | 312; 312 Patients with or without CMV DNAemia
Completed | 144; 144 Patients with or without CMV DNAemia | 422; 422 Patients with or without CMV DNAemia | 312; 312 Patients with or without CMV DNAemia
Not Completed | 0; 0 Patients with or without CMV DNAemia | 0; 0 Patients with or without CMV DNAemia | 0; 0 Patients with or without CMV DNAemia

BASELINE CHARACTERISTICS:
Groups:
- Pre-CMV DNAemia: Patients with CMV DNAemia detected prior neutrophil's engraftment
- No CMV: Patients without CMV DNAemia
- Total: Total of all reporting groups
Arm/Group | Pre-CMV DNAemia | Post-CMV DNAemia | No CMV | Total
Number analyzed (Participants) | 144 | 422 | 312 | 878
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 134 | 370 | 275 | 779
  >=65 years | 10 | 52 | 37 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 174 | 135 | 366
  Male | 87 | 248 | 177 | 512
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 144 | 422 | 312 | 878
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Engraftment (Days) Stratified by CMV DNaemia Occurring Before or After Neutrophil's Engraftment
Description: absolute neutrophil count ≥500/mm3 on 3 consecutive days,, the first of which being time of engraftment.
Time Frame: 30 days
Population: Patients with CMV DNAemia
Measure: Median (Full Range); unit: days
Groups:
- Pre-CMV DNAemia: episodes of CMV DNAemia that were detected prior to engraftment
- Post-CMV DNAemia: episodes of CMV DNAemia that were detected after engraftment
Arm/Group | Pre-CMV DNAemia | Post-CMV DNAemia
Number analyzed (Participants) | 144 | 422
days | 17 [8 to 42] | 19 [5 to 57]

2. Secondary Outcome: Overall Mortality
Description: total number of deaths from any cause
Time Frame: 1 year
Population: Patients with CMV DNAemia detected prior or after neutrophil's engraftment
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-CMV DNAemia | Post-CMV DNAemia
Number analyzed (Participants) | 144 | 422
Participants | 54 | 131

3. Secondary Outcome: Non-relapse Mortality
Description: total number of deaths without relapse or underlying disease progression
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-CMV DNAemia | Post-CMV DNAemia
Number analyzed (Participants) | 144 | 422
Participants | 34 | 96

ADVERSE EVENTS:
Time Frame: 1 year
Description: death from any cause
Groups:
- No CMV DNAemia: Patients without CMV DNAemia
Arm/Group | Pre-CMV DNAemia | Post-CMV DNAemia | No CMV DNAemia
All-Cause Mortality (participants affected / at risk) | 54/144 | 131/422 | 94/312
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/422 | 0/312
Other Adverse Events (participants affected / at risk) | 0/144 | 0/422 | 0/312

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03889028/Prot_SAP_000.pdf